CLINICAL TRIAL: NCT06406842
Title: Perioperative Application of Hemodynamic Management Based on Regional Cerebral Oxygen Saturation Monitoring of Cerebral Autoregulation in Carotid Endarterectomy
Brief Title: Association Between Local Cerebral Oxygenation Monitoring and Postoperative Stroke in Carotid Endarterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202422047
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Carotid Endarterectomy; Cerebral Autoregulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigator of control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The autoregulation group (Experimental): In the autoregulation group, anesthesiologist will maintain that the cerebral oxygen index value below 0.3. If cerebral oxygen index exceeds the threshold, Norepinephrine or Phenylephrine will be infused continuously, or arterial partial pressure of oxygen or arterial partial pressure of carbon dioxide will be adjusted to increase regional cerebral oxygen saturation.
  Interventions: Other: Cerebral oxygenation index guided hemodynamics management
- The routine group (No Intervention): In the routine group, the screen of the collection monitor will be covered by a black cloth . Anesthesiologist will not have access to the patient's cerebral oxygen index value. Anesthesiologist will strive to maintain mean arterial pressure within a ± 20% range of their baseline mean arterial pressure. Outside of this range, the same vasoactive drugs will be employed for modulation. Additionally, anaesthesiologists will maintain PaCO₂ within the range of 35-45 mmHg and set the fraction of inspired oxygen at 50%.

INTERVENTIONS:
Other: Cerebral oxygenation index guided hemodynamics management — In the autoregulation group, anesthesiologist will maintain that the cerebral oxygen index value below 0.3. If cerebral oxygen index exceeds the threshold, norepinephrine or phenylephrine will be infused continuously, or arterial partial pressure of oxygen or arterial partial pressure of carbon dioxide will be adjusted to increase regional cerebral oxygen saturation.
  Arms: The autoregulation group

SUMMARY:
Carotid endarterectomy (CEA) is used to treat symptomatic extracranial internal carotid artery stenosis. The occult stroke of CEA patients evaluated by magnetic resonance imaging 3 days after operation was as high as 17%. Cerebral blood flow autoregulation (CA) is the ability of the brain to maintain the relative stability of cerebral blood flow, and cerebral oxygen index (COx) can be used to reflect CA. A negative value of cerebral oxygen index or a value near zero indicates that CA is complete, and cerebral oxygen index close to 1 indicates that CA has lost its ability. In theory, real-time monitoring of CA function by cerebral oxygen index and individualized management strategy with this goal can potentially reduce perioperative ischemic brain injury. The purpose of this study is to explore the influence of the management strategy of monitoring CA function based on regional cerebral oxygen saturation on the postoperative neurological complications of CEA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective carotid endarterectomy
* ASA Ⅱ or Ⅲ
* aged 18-80 years old

Exclusion Criteria:

* preoperative moderate and severe cognitive impairment
* preoperative psychotropic medication history within one year
* history of neurosurgery
* have speech or language impairments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative cerebral ischemic events | postoperative 3 day
  Our primary outcome will be the incidence of new ischemic brain injury within 3 days after surgery, defined as new infarct focus detected by magnetic resonance imaging diffusion-weighted imaging or computed tomography, with or without new-onset limb weakness, paresthesia, or language abnormalities. Diffusion-weighted imaging sequences will be used at each scan to detect acute ischemic brain lesions.

SECONDARY OUTCOMES:
The incidence of postoperative delirium | The first 3 days after surgery
  The incidence and severity of postoperative delirium will be assessed during the first 3 days after surgery. Delirium will be assessed twice daily between 8:00-10:00 and 18:00-20:00 in ward patients with the Richmond Agitation Sedation Scale (RASS) and the 3 min diagnostic interview for CAM (3D-CAM). ICU patients will be similarly assessed with RASS and the confusion assessment method for ICU (CAM-ICU). Any positive 3D-CAM or CAM-ICU assessment will be considered evidence of delirium.
Basic Cognition Assessment | The day before surgery and postoperative day 4 or 5
  Postoperative basic cognitive function will be assessed by Mini-mental State Examination. This will be rated on a scale from 0 to 30, higher cores corresponded to higher levels of cognitive function.
Advanced Cognitive Assessment | The day before surgery and postoperative day 4 or 5
  Postoperative basic cognitive function will be assessed by Montreal Cognitive Assessment-Basic Examination. This will be rated on a scale from 0 to 30, higher cores corresponded to higher levels of cognitive function.
Pain assessment | At 24, 48, and 72 hours post-surgery
  Pain scores will be recorded at rest and during movement . The pain was rated on a scale from 0 to 10, where 0 indicated no pain and 10 indicated the worst possible pain. Higher scores corresponded to higher levels of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming MD Peng, Ph.D, Principal Investigator — Beijing Tian Tan Hospital
Locations (2):
- China (2):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li M, Yin X, Liang C, Tao C, Yan Q, Zeng M, Li S, Sessler DI, Wang R, Zhao L, Peng Y. Effect of perioperative haemodynamic management based on cerebral autoregulation monitored by Cerebral Oximetry Index during carotid endarterectomy: protocol of a randomised trial. BMJ Open. 2025 Jun 19;15(6):e094156. doi: 10.1136/bmjopen-2024-094156. PMID 40537236